CLINICAL TRIAL: NCT05082662
Title: Randomized,Fully-replicated,Single Oral Dose,Open-label,Crossover BE Study to Compare Diclofenac Potassium Coated Tablet (50 mg Diclofenac Potassium) Versus Cataflam® 50 Coated Tablet (50 mg Diclofenac Potassium) in Healthy Subjects in Fasting State
Brief Title: Bioequivalence Study to Compare Diclofenac Potassium Coated Tablet Versus Cataflam® 50 Coated Tablet
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 974-2020
Record Dates: First submitted 2021-09-14; First posted 2021-10-19 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Non-steroidal Anti-inflammatory (NSAID); Analgesic; Antipyretic
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac Potassium coated tablet (50 mg Diclofenac Potassium) (Experimental)
  Interventions: Drug: Diclofenac Potassium coated tablet (50 mg Diclofenac Potassium); Drug: Cataflam® 50 coated tablet
- Cataflam® 50 coated tablet (50 mg Diclofenac Potassium) (Active Comparator)
  Interventions: Drug: Diclofenac Potassium coated tablet (50 mg Diclofenac Potassium); Drug: Cataflam® 50 coated tablet

INTERVENTIONS:
Drug: Diclofenac Potassium coated tablet (50 mg Diclofenac Potassium) — One Diclofenac tablet was administered orally.
Drug: Cataflam® 50 coated tablet — One Diclofenac tablet was administered orally.

SUMMARY:
Randomized, four-way, four-period, fully-replicated, single oral dose, open-label, crossover, bioequivalence study to compare Diclofenac Potassium coated tablet (50 mg Diclofenac Potassium) versus Cataflam® 50 coated tablet (50 mg Diclofenac Potassium), in healthy subjects under fasting condition

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged between eighteen & fifty years (18 - 50).
* The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, vital signs, physical examination & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for hepatitis (B & C) viruses and Human Immunodeficiency Virus (HIV).
* There is no evidence of psychiatric disorder, antagonistic personality and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* For female subjects: negative pregnancy test and the woman is using two reliable contraception methods.
* The subject has normal gastrointestinal, cardiovascular system and ECG recording.
* The subject kidney and liver (AST & ALT enzymes) functions tests are within normal range.

Exclusion Criteria:

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is vegetarian.
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 10 hours after dosing in all study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
* The subject has consumed drugs that may affect pharmacological or pharmacokinetic properties (Voriconazole and Aspirin) two weeks before dosing, during the study and two weeks after dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 10 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for Cmax
AUC0-t | 10 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for AUC0-t
AUC0-∞ | 10 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for AUC0-∞

SECONDARY OUTCOMES:
Tmax | 10 hours
  The descriptive statistics including Maximum, Minimum and Median values will be measured for Tmax
Thalf | 10 hours
  Thalf was calculated from 0.693/ λz
Kelimination | 10 hours
  The terminal elimination rate constant (Kelimination or λz) was estimated for each subject and for each treatment via linear regression of the last points (at least three points will be used) at the terminal phase of the log-concentration versus time curve of each subject
Blood pressure (safety and tolerability) | At pre-dosing, 2, 4, 6, 8, and 10 hours post dosing, ± 45 minutes of scheduled time
  Clinically significant abnormal deviations. Normal range of blood pressure > 90/60 and <140/90 mmHg.
Pulse (safety and tolerability) | At pre-dosing, 2, 4, 6, 8, and 10 hours post dosing, ± 45 minutes of scheduled time
  Clinically significant abnormal deviations. Normal range of Pulse 60-100 bpm.
Temperature(safety and tolerability) | At pre-dosing; 4, and 10 hours post dosing, ± 45 minutes of scheduled time
  Clinically significant abnormal deviations. Normal range of temperature 36.5-37.5 ºC.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- ACDIMA Biocenter, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided